CLINICAL TRIAL: NCT03503539
Title: Are the Stone Density and Location Useful Parameters That Can Determine the Endourological Surgical Technique for Kidney Stones That Are Smaller Than 2 cm? Prospective Randomized Controlled Trial
Brief Title: Are the Stone Density and Location Useful Parameters for Small Kidney Stones?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Adnan Gucuk, Associate Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AbantIBU-AG001
Record Dates: First submitted 2018-03-28; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Kidney Calculi; Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mini percutaneous nephrolithotomy (Experimental): All operations were performed or supervised by the same surgeon. Right after the patients in mini-PNL group were placed a 5F ureteral catheter with general anesthesia, they were had a prone position and the access was performed by choosing the optimal calyx to reach the stone following the contrast agent was given. The guide wire was then placed and the stones were broken with a laser lithotripter using a 12F nephroscope (Modular minimally invasive PCNL system, Karl Storz, Tuttlingen, Germany) following the dilatation using an one step dilator with a 16.5F access sheath. When necessary, stones were removed using the stone removal forceps. Right after a 14-Fr nephrostomy tube was inserted and an antegrade pyelography was taken, the operation was terminated.
  Interventions: Procedure: Mini percutaneous nephrolithotomy
- Retrograde intrarenal surgery (Active Comparator): Following the general anesthesia performed, a safety guide wire was placed and semirigid ureteroscopy (9.5 / 11.5F) was performed. Stones were fragmented using a 270 micron meter laser fiber with the help of 7.5-F fiber optic flexible ureterorenoscope after the placement of ureteral access sheat (9.5 / 11.5 F). Stone fragmentation was accomplished using a laser energy of 0.5-1.5 J and a rate of 5-15 Hz and adjusting this range according to stone hardness. 4.7F JJ stent was routinely placed at the end of the operation because of worries about possible edema etc. due to access sheath. In this group, access sheath could not be placed in 2 patients due to the small diameter of the ureter, and JJ stent was placed, and 2 weeks later, the procedure was performed as it was in the others.
  Interventions: Procedure: Retrograde intrarenal surgery

INTERVENTIONS:
Procedure: Mini percutaneous nephrolithotomy
  Arms: Mini percutaneous nephrolithotomy
Procedure: Retrograde intrarenal surgery
  Arms: Retrograde intrarenal surgery

SUMMARY:
The investigators aimed to evaluate whether these parameters could be guides for us in the selection of RIRS or Mini-PNL procedures in kidney stones that are smaller than 2 cm.

The patients that have kidney stones smaller than two cm and be planned to undergo surgery were randomized into 2 groups prospectively. RIRS was performed in the RIRS group using a 7.5-F fiberoptic flexible ureterorenoscope while Mini-PCNL group was dilated up to 16.5F and mini-PCNL was performed with 12F nephroscopy. Preoperative characteristics, operative and postoperative results were compared in two groups. Thereafter, intra and intergroup comparisons were made to determine the effects of HU value, indicating the stone density, higher or less than 677 and the stone location on stone-free rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients were evaluated with non-contrast abdominopelvic CT after a detailed anamnesis and physical examination.
* Patients, who had a kidney stone with a maximum diameter of less than 2 cm and who did not prefer to undergo ESWL, were taken into the study.

Exclusion Criteria:

* Patients with anomalous kidneys, skeletal deformities, severe obesity (BMI> 35) and those underwent ESWL treatment previously for the same stone were excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Stone free rate | 1 year
  Stone-free conditions were determined by low-dose spiral CT taken in postoperative third month

SECONDARY OUTCOMES:
Mean fluoroscopy time | İntraoperative duration of flouroscopy
  İntraoperative duration of flouroscopy time

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Demirbas A, Resorlu B, Sunay MM, Karakan T, Karagoz MA, Doluoglu OG. Which Should be Preferred for Moderate-Size Kidney Stones? Ultramini Percutaneous Nephrolithotomy or Retrograde Intrarenal Surgery? J Endourol. 2016 Dec;30(12):1285-1289. doi: 10.1089/end.2016.0370. PMID 27706948
- [Result] Jacquemet B, Martin L, Pastori J, Bailly V, Guichard G, Bernardini S, Chabannes E, Bittard H, Kleinclauss F. Comparison of the efficacy and morbidity of flexible ureterorenoscopy for lower pole stones compared with other renal locations. J Endourol. 2014 Oct;28(10):1183-7. doi: 10.1089/end.2014.0286. Epub 2014 Sep 12. PMID 24811281
- [Result] Resorlu B, Unsal A, Gulec H, Oztuna D. A new scoring system for predicting stone-free rate after retrograde intrarenal surgery: the "resorlu-unsal stone score". Urology. 2012 Sep;80(3):512-8. doi: 10.1016/j.urology.2012.02.072. Epub 2012 Jul 26. PMID 22840867
- [Result] Resorlu B, Oguz U, Resorlu EB, Oztuna D, Unsal A. The impact of pelvicaliceal anatomy on the success of retrograde intrarenal surgery in patients with lower pole renal stones. Urology. 2012 Jan;79(1):61-6. doi: 10.1016/j.urology.2011.06.031. PMID 21855968
- [Result] Turk C, Petrik A, Sarica K, Seitz C, Skolarikos A, Straub M, Knoll T. EAU Guidelines on Diagnosis and Conservative Management of Urolithiasis. Eur Urol. 2016 Mar;69(3):468-74. doi: 10.1016/j.eururo.2015.07.040. Epub 2015 Aug 28. PMID 26318710
- [Result] Gucuk A, Uyeturk U, Ozturk U, Kemahli E, Yildiz M, Metin A. Does the Hounsfield unit value determined by computed tomography predict the outcome of percutaneous nephrolithotomy? J Endourol. 2012 Jul;26(7):792-6. doi: 10.1089/end.2011.0518. Epub 2012 Feb 10. PMID 22201298